CLINICAL TRIAL: NCT01173887
Title: Multicenter, Randomized, Open-label, Parallel-group Study to Compare mLSG15 + KW-0761 to mLSG15 in Subjects With CCR4-positive Adult T-cell Leukemia-lymphoma (Untreated Primary Disease)
Brief Title: Multicenter, Randomized, Open-label, Parallel-group Study to Compare mLSG15 + KW-0761 to mLSG15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0761-003
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Adult T-cell Leukemia-Lymphoma
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell | interventions — mogamulizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mLSG15 (Active Comparator)
  Interventions: Drug: VCAP/AMP/VECP(mLSG15)
- mLSG15 + KW-0761 (Experimental)
  Interventions: Biological: KW-0761

INTERVENTIONS:
Drug: VCAP/AMP/VECP(mLSG15) — VCAP(Vincristine Sulfate, Cyclophosphamide Hydrate, Doxorubicin Hydrochloride, Prednisolone); AMP(Doxorubicin Hydrochloride, Ranimustine, Prednisolone); VECP(Vindesine Sulfate, Etoposide, Carboplatin, Prednisolone)
  Arms: mLSG15
Biological: KW-0761 — VCAP/AMP/VECP(mLSG15) + KW-0761
  Arms: mLSG15 + KW-0761

SUMMARY:
This is a multicenter, randomized, open-label, parallel-group study to compare mLSG15 + KW-0761 to mLSG15 in subjects with CCR4-positive adult T-cell leukemia-lymphoma (untreated primary disease). The primary variable is an efficacy of KW-0761 used as an add-on therapy to mLSG15 as measured in terms of complete response rate (CR/CRu) in the best overall response assessment for antitumor effect. The secondary variables include response rate (CR/CRu/PR) in the best overall response assessment for antitumor effect, complete or response rates by lesion site in the best overall response assessment for antitumor effect, progression-free survival and overall survival. The safety and pharmacokinetic profiles of KW-0761 will be also determined.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been positive for serum anti-human T-cell lymphotropic virus type I antibody
* Subjects with hematologically or pathohistologically confirmed as peripheral lymphoid tumor which surface antigen analysis has identified to be of T-cell origin
* Subjects who have been classified into acute subtype, the lymphoma subtype or chronic subtype with poor prognostic factors
* Subjects who have been positive for CCR4 by CCR4 expression analysis
* Subjects who have never been treated for adult T-cell leukemia-lymphoma
* Subjects who have presented enlarged lymph nodes, tumor nodules in extranodal organs, abnormal lymphocytes in peripheral blood or cutaneous lesions
* Subjects with a performance status of 0 to 2
* Subjects who have been negative for HBs antigen and anti-HCV antibody
* Subjects who have given written voluntary informed consent to participate in the study

Exclusion Criteria:

* Subjects who are scheduled for transplant therapy such as hematopoietic stem-cell transplantation
* Subjects who had myocardial infarction within 12 months before study enrollment or who have cardiac disease that may worsen during treatment with doxorubicin
* Subjects who have been positive for anti-HIV antibody
* Subjects with active multiple cancer
* Subjects with a history of allergic reactions to therapeutic antibodies
* Subjects who require emergency radiotherapy for treating the symptoms caused by bulky masses or who may require such radiotherapy after the start of the study
* Subjects who are pregnant, lactating or of childbearing potential, or who are planning to have children

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Complete response rate in the best overall response assessment for antitumor effect | After cycle 2 and cycle 4

SECONDARY OUTCOMES:
Response rate in the best overall response assessment for antitumor effect, complete or response rates by lesion site in the best overall response assessment for antitumor effect | After cycle 2 and cycle 4.
Progression-free survival and Overall survival | During the study period at least once every two months in the first year and once every three months in the second and subsequent years.
Adverse events | During the study period
anti-KW-0761 antibody | Before 1st and 5th dosing, 14 days after 8th or last dosing and at the start of post-treatment.
Plasma KW-0761 concentrations and pharmacokinetic parameters | Before and after 1st, 2nd, 3rd, 4th, 5th, 6th, 7th and 8th dosing, 14 days after 8th or last dosing, and at the start of post-treatment.

CONTACTS AND LOCATIONS:
Locations (19):
- Japan (19):
  - Fukuoka University Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - National Kyushu Cancer Center, Fukuoka
  - Imamura Bun-in Hospital, Kagoshima
  - Kagoshima University Hospital, Kagoshima
  - Kokura Memorial Hospital, Kitakyushu
  - Kumamoto University Hospital, Kumamoto
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - NTT West Japan Kyushu Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Aichi Cancer Center Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Heartlife Hospital, Okinawa
  - Oita Prefectural Hospital, Ōita
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - Sasebo City General Hospital, Sasebo
  - National Cancer Center Hospital, Tokyo
  - Ehime University Hospital, Tōon

REFERENCES:
- [Derived] Ishida T, Jo T, Takemoto S, Suzushima H, Uozumi K, Yamamoto K, Uike N, Saburi Y, Nosaka K, Utsunomiya A, Tobinai K, Fujiwara H, Ishitsuka K, Yoshida S, Taira N, Moriuchi Y, Imada K, Miyamoto T, Akinaga S, Tomonaga M, Ueda R. Dose-intensified chemotherapy alone or in combination with mogamulizumab in newly diagnosed aggressive adult T-cell leukaemia-lymphoma: a randomized phase II study. Br J Haematol. 2015 Jun;169(5):672-82. doi: 10.1111/bjh.13338. Epub 2015 Mar 2. PMID 25733162